CLINICAL TRIAL: NCT04673630
Title: A Phase I, Open-label Study to Evaluate the Pharmacokinetics of Tezepelumab in Children ≥ 5 to 11 Years of Age With Mild, Moderate, or Severe Asthma (TRAILHEAD)
Brief Title: Study to Evaluate the Pharmacokinetics of Tezepelumab in Children With Asthma
Acronym: TRAILHEAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5180C00025
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: Mild asthma; Moderate asthma; Severe asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Masking Description: No masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — Single dose subcutaneous injection

SUMMARY:
This study will evaluate the pharmacokinetic (PK) profile of a single subcutaneous (SC) dose of tezepelumab in children aged ≥ 5 to 11 years with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and written informed assent and any locally required authorisation obtained from the subject and legal representative prior to any study related procedure taking place.
* Age 5 to 11 years (inclusive) at Visit 1 and Visit 2 (Day 1). Type of Subject and Disease Characteristics
* Documented physician diagnosed asthma for at least 6 months prior to Visit 1.
* Documented treatment with total daily dose of either low, medium, or high dose ICS for at least 6 months, as described in Step 2 to Step 4 of GINA guidelines (GINA 2020) with stable dose for at least 3 months prior to Visit 1.
* Pre bronchodilator (BD) FEV1 of ≥ 50% of predicted normal value at Visit 1
* Body weight ≥ 16 kg at Visit 1 and Visit 2 (Day 1).

Exclusion Criteria:

* History of any clinically significant disease or disorder other than asthma which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History of a deterioration in asthma or asthma exacerbation that required a burst of systemic corticosteroids within 6 weeks of Visit 1, up to and including Visit 2 (Day 1).
* History of hospitalisation (overnight admission) for asthma within 3 months of Visit 1, up to and including Visit 2 (Day 1).
* History of a life threatening asthma exacerbation requiring intubation or mechanical ventilation.
* History of systemic corticosteroid use for the maintenance treatment of asthma within 6 weeks of Visit 1, up to and including Visit 2 (Day 1) and discouraged until EOS.
* History of cancer.
* History of hypersensitivity or anaphylactic reaction to any biologic therapy.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grigg, MD, Principal Investigator — Royal London Hospital, United Kingdom
Locations (5):
- Research Site, Budapest, Hungary
- Research Site, Cape Town, South Africa
- United Kingdom (3):
  - Research Site, Bristol
  - Research Site, Glasgow
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00025&attachmentIdentifier=4e88e9dc-f504-4df4-ab92-5048a89f274c&fileName=D5180C00025_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I open-label study was conducted in pediatric participants with mild, moderate, or severe asthma at 6 investigational sites in the UK, Hungary, and South Africa between 23 February 2021 and 27 September 2022.
Pre-assignment Details: This study consists a screening period (14 days), and a single dose treatment (Day 1) and follow-up period (85 days). A total of 18 participants were treated in the study.
Groups:
- Tezepelumab: Participants received a single dose of tezepelumab subcutaneous (SC) injection on Day 1.
Period: Overall Study
Arm/Group | Tezepelumab
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all participants who received at least 1 dose of tezepelumab.
Groups:
- Tezepelumab: Participants received a single dose of tezepelumab SC injection on Day 1.
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 1
  White | 6
  Other | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Tezepelumab
Description: Blood samples were collected to determine the Cmax of tezepelumab. The Pharmacokinetic (PK) parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: The PK analysis set included participants in the Safety Analysis set that had at least 1 detectable tezepelumab serum concentration from a sample collected postdose that was assumed not to be affected by factors such as important protocol deviations (eg, incorrect dose of study drug received).
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
microgram per milliliter (mcg/mL) | 27.1 (11.9)

2. Primary Outcome: Time to Achieve Maximum Observed Serum Concentration (Tmax) of Tezepelumab
Description: Blood samples were collected to determine the tmax of tezepelumab. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
day | 3.47 [1.92 to 9.96]

3. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero to The Last Measurable Concentration (AUC0-last) of Tezepelumab
Description: Blood samples were collected to determine the AUC0-last of tezepelumab and calculated by linear up/log down trapezoidal summation. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
day*mcg/mL | 872 (285)

4. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Tezepelumab
Description: Blood samples were collected to determine the AUC0-inf of tezepelumab and calculated by linear up/log down trapezoidal summation and extrapolated to infinity by the addition of the last quantifiable concentration divided by the terminal rate constant. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
day*mcg/mL | 974 (320)

5. Primary Outcome: Terminal Phase Elimination Half-Life (t1/2) of Tezepelumab
Description: Blood samples were collected to determine the t1/2 of tezepelumab and calculated as ln(2)/λZ, where λZ is the first-order rate constant associated with the terminal (log-linear) elimination phase. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
day | 25.7 (5.94)

6. Primary Outcome: Apparent Clearance (CL/F) of Tezepelumab
Description: Blood samples were collected to determine the CL/F of tezepelumab and estimated as dose divided by AUC0-inf. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter per day
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
liter per day | 0.0802 (0.0295)

7. Primary Outcome: Apparent Steady-State Volume of Distribution (Vss/F) of Tezepelumab
Description: Blood samples were collected to determine the Vss/F of tezepelumab and estimated as CL/F*mean residence time (MRT), where MRT=Area under the moment curve of the analyte in the sampled matrix from zero (predose) extrapolated to infinite time/(AUC0-inf). The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
liter | 3.08 (1.32)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Tezepelumab
Description: Blood samples were collected to determine the Vz/F of tezepelumab and estimated as CL/F*1/ λZ. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 3, 7, 11, 15, 29, 57 and 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
liter | 2.98 (1.26)

9. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Tezepelumab
Description: Blood samples were analyzed for the presence of ADAs for tezepelumab using validated assays. ADA prevalence was defined as ADA positive at baseline and/or post baseline. ADA incidence was defined as the percentage of treatment-emergent ADA positive participants in a population. Treatment induced ADA positive was defined as ADA negative at baseline and post-baseline ADA positive. Treatment-boosted ADA positive was defined as baseline positive ADA titre that was boosted to a 4-fold or higher level following study drug administration. Treatment-emergent ADA positive was defined as either treatment-induced ADA positive or treatment-boosted ADA positive.
Time Frame: Predose and within ± 1 hour of postdose on Day 1; on Days 29 and 85
Population: The Safety analysis set included all participants who received at least 1 dose of tezepelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab
Number analyzed (Participants) | 18
Participants
  ADA prevalence | 3
  Only baseline ADA positive | 2
  Baseline and at least 1 post-baseline ADA positive | 1
  Baseline ADA positive regardless of post-baseline | 3
  Any post-baseline ADA positive | 1
  Treatment-induced ADA positive | 0
  Treatment-boosted ADA positive | 0
  Treatment-emergent ADA positive | 0

ADVERSE EVENTS:
Time Frame: From the first dose administration (Day 1) up to study completion (End of Study/Day 85 visit) or withdrawal date
Description: The Safety analysis set included all participants who received at least 1 dose of tezepelumab.
Arm/Group | Tezepelumab
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 7/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=18)
COVID-19 (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT04673630/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04673630/SAP_001.pdf